CLINICAL TRIAL: NCT03970187
Title: Randomized Controlled Trial on the Efficacy of a VR Exposure-based Eye Contact Training‬ to Reduce Fear of Public Speaking
Brief Title: Investigation of the Efficacy of a VR Exposure-based Eye Contact Training‬ to Reduce Fear of Public Speaking
Acronym: ASSIST-2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division of Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-00514
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Fear of Public Speaking (Subclinical)
MeSH Terms: conditions — Glossophobia

STUDY DESIGN:
Intervention Model Description: Randomized controlled single-blind study design.
Who Masked: Investigator
Masking Description: Investigators evaluating the (external) performance in the in vivo Public Speech Test (PST) will be blinded (unaware of group assignment of participants, single-blind).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure (Experimental): Phase 1 (visit 1): 60 minutes exposure-based eye contact training in VR Phase 2 (home training): 9 blocks of 20 minutes exposure-based eye contact training in VR, distributed over a total duration of maximally 2 weeks
  Interventions: Other: Exposure-based eye contact training in Virtual Reality (VR)
- Control (No Intervention): Phase 1 (visit 1): waitlist. In order to prevent systematic preparation for the subsequent PST, a 60 minutes virtual reality games with fear-unrelated content will serve as the control intervention.
  Phase 2 (home training): waitlist

INTERVENTIONS:
Other: Exposure-based eye contact training in Virtual Reality (VR) — The intervention is an App for virtual reality. The VR App provides three different virtual scenarios. Participants will be asked to stand in front of a virtual audience and to maintain eye contact with audience members. The advance to higher difficulty levels is according to a pre-defined exposure scheme. Participants will be given all instructions via the App.
  There will be three sessions on one day (duration of 20 min each) in study phase 1. The indication is disproportionate fear of being evaluated by others and reduced eye contact as a typical avoidance strategy in individuals with fear of public speaking. In the study phase 2, there will be nine sessions spanning over two weeks (duration of 20 min each, with maximally one session per day). The indication is disproportionate fear of being evaluated by others and reduced eye contact as a typical avoidance strategy in individuals with fear of public speaking.
  Arms: Exposure

SUMMARY:
Investigation of the efficacy of an eye contact training App in virtual reality, based on principles of exposure therapy for the treatment for subjects with fear of public speaking.

DETAILED DESCRIPTION:
The study will be conducted as a randomized controlled single-blind study in a parallel groups design.

Participants will be divided into groups afraid of public speaking with and without fulfilling the criteria of social anxiety (according to DSM-V), which can represent a clinically relevant and more generalized form of public speaking anxiety. The treatment for the participants solely differs in terms of whether they receive (1) the VR exposure or (2) a fear-unrelated VR task (study phase 1) or no treatment at all (study phase 2), resulting in the following 2 groups:

* Group 1 (treatment group) consists of individuals with fear of public speaking that will (in study phase 1) receive a three-session VR exposure and undergo (in study phase 2) a 2-week treatment period with the same VR scenarios, each repeated three times.
* Group 2 (control group) consists of individuals with fear of public speaking that will not receive any active treatment but complete a distractor task in VR in study phase 1 and no treatment in study phase 2.

In study phase 1, the treatment group receives three VR exposure sessions each lasting for 20 minutes, whereas the control group completes three virtual distractor tasks (e.g. virtual tours) of identical duration. In study phase 2, the treatment group completes a home training spanning two weeks (9 x 20-minutes sessions), whereas the control group does not receive any treatment (untreated comparison group).

In study phase 1, before and after the virtual exposure session, participants undergo an in vivo PST to assess the acute effects of the VR exposure-based eye contact training App.

In study phase 2, the participants undergo a third in vivo PST to assess the training effects of the VR exposure-based eye contact training after two weeks of home training.

This design allows a direct isolation and comparison of acute effects (study phase 1) and of training effects (study phase 2) and therefore enables an overall estimation of the effectiveness of the VR exposure-based eye contact training.

Approximately 96 participants between 18 and 40 years with fear of public speaking will take part in the study. Approximately 1 to 5 weeks after having finished the first study phase, all participants that have not dropped out will take part in the second study phase.

ELIGIBILITY:
Inclusion Criteria:

* Fear of public speaking, assessed by two separate aspects:
* High fear in social situations including the potential of being evaluated by others
* Social situations can only be withstood under high fear or are avoided
* Aged between 18-40
* Fluent in German

Exclusion Criteria:

* BDI-II sumscore >= 20
* Suicidal ideation (BDI-II item 9 > 0)
* Serious medical or psychological condition, other than social anxiety (including Depression, Epilepsy and Migraine)
* Concurrent psychotherapy
* Previous exposure-based therapy for social anxiety (including public speaking anxiety) or other anxiety disorders
* Parallel participation in another psychological or medical study
* Chronic medication intake (except oral contraceptives)
* Chronic drug intake (i.e. LSD, mushrooms, Ecstasy, MDMA, amphetamines etc.)
* Medication intake before visits (less than 24 h)
* Alcohol intake before visits (less than 12 h)
* Cannabis or other psychoactive substances (including benzodiazepines) intake before visits (less than 5 days)
* Restricted 3D sight
* For women: Current pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS, fear) | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Fear of public speaking is quantified by means of SUDS-ratings during a Public Speaking Test (PST) in vivo.

SECONDARY OUTCOMES:
Global external assessment of performance in an in vivo public speech test | Assessing change between baseline and predefined follow-up time points during 11 weeks
  The global external assessment of performance is done by averaging VAS-ratings (range from 0 = very bad performance to 100 = very good performance) of the PST from three independent members of a committee (experimenters) and a forth experimenter that will rate the performances using a video and audio recording from the speeches.
Total time of eye contact during an in vivo public speech test | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Total time of eye contact is measured by a mobile eye tracking device from Pupil Labs and operationalized by the number of frames the gaze is in predefined regions of interest comprising the eyes of the committee members.
Fear of eye contact (SUDS, eye contact) | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Fear of public speaking is quantified by means of SUDS-ratings during a Public Speaking Test (PST) in vivo.
Global self-assessment of performance in an in vivo public speech test | Assessing change between baseline and predefined follow-up time points during 11 weeks
  The global self-assessment of performance is done by a VAS-ratings (range from 0 = very bad performance to 100 = very good performance) of the PST
Global subjectively perceived improvement of fear, eye contact and performance after single VR-exposure/waitlist | Assessed at visit 1 after completing the second PST
  Global subjectively perceived improvement of fear, eye contact and performance by the VR eye contact training App will be done by VAS-ratings
Global subjectively perceived improvement of fear, eye contact and performance after VR-training/waitlist | Assessed at visit 2 after completing the PST
  Global subjectively perceived improvement of fear, eye contact and performance by the VR eye contact training App will be done by VAS-ratings
Questionnaire for social anxiety (Soziale-Phobie-Inventar; SPIN) | Assessing change between baseline and predefined follow-up time points during 11 weeks
  The SPIN is a 17-item questionnaire developed by the Psychiatry and Behavioral Sciences Department at Duke University. It is effective in screening for, and measuring the severity of fear related to the negative evaluation by others. The 17 items cover different aspects of the anxiety such as fear, avoidance, and physiological symptoms on 5-point Likert scales. The statements of the SPIN items indicate the particular signs of public speaking anxiety (e.g. "I am bothered by blushing in front of people"). The SPIN demonstrates solid psychometric properties and is valid as a measurement for the severity and clinical relevance of fear related symptoms (Connor et al., 2000).
Questionnaire for fear of negative evaluation (The Furcht vor negativer Evaluation - Kurzskala; FNE-K) | Assessing change between baseline and predefined follow-up time points during 11 weeks
  The FNE-K is a frequently used, valid, and reliable self-report questionnaire consisting of 12 items measuring fear and distress related to negative evaluation by others (e.g. "I am afraid that people will find fault with me") on 4-point Likert scales. The FNE-K has demonstrated good reliability and validity (Reichenberger et al., 2016).
Eye-tracking measures | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Gaze behaviour (fixation frequency and location, scan path characteristics) and pupil size
Physiological measures | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Salivary cortisol levels

OTHER OUTCOMES:
Feature-specific external and self-assessment of performance in an in vivo public speech test (VAS-ratings) | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Feature-specific assessment of the participants performance in the in vivo PST is measured by VAS-ratings (from 0 = very bad to 100 = very good) from three independent members of a committee. A forth experimenter will rate the performances using a video and audio recording from the speeches. 8 specific VAS-ratings covering nonverbal aspects of performances (e.g. facial expression, gestures etc.) are divided into two subscales with 4 VAS-ratings each (1 = speech, 2 = appearance).
Vocal indices of stress | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Vocal indices of stress comprise f.e. level and variability of the fundamental frequency or the active speech duration. They will be measured by analysing the audio recordings during the PST.
Simulation sickness in VR | Assessing change between baseline and predefined follow-up time points during 11 weeks
  Safety outcome, assessed by the Simulator Sickness Questionnaire (SSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, MD, Study Director — University of Basel, Division of Cognitive Neuroscience
Locations (1):
- University of Basel, Division of Cognitive Neuroscience, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No